CLINICAL TRIAL: NCT03747315
Title: Assessment of a Functional Test to Detect Familial Mediterranean Fever
Brief Title: A Diagnostic Test for Familial Mediterranean Fever
Acronym: DEPIST-FMF
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0710
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Familial Mediterranean Fever (patients): Patients with previously confirmed Familial Mediterranean Fever (based on clinical criteria)
  Interventions: Other: In vitro functional test
- Control group (patients): Patients with symptoms similar to that of Familial Mediterranean Fever (e.g. Behcet disease, Crohn, sepsis..) but without confirmed Familial Mediterranean Fever.
  Interventions: Other: In vitro functional test
- Healthy donors: Patients without symptoms (anonymous blood donors)
  Interventions: Other: In vitro functional test

INTERVENTIONS:
Other: In vitro functional test — Measurement of interleukin-1beta secretion by monocytes and measurement of cell death upon Pyrin inflammasome activation by kinase inhibitor on an additional blood sample (4 ml for children under 12 and 10 ml for children 12 years and older and adults) during a sample for patient care.
  Groups: Control group (patients); Familial Mediterranean Fever (patients)
Other: In vitro functional test — Measurement of interleukin-1beta secretion by monocytes and measurement of cell death upon Pyrin inflammasome activation by kinase inhibitor on samples from healthy subjects who donated their blood to the French Blood Establishment.
  Groups: Healthy donors

SUMMARY:
Familial Mediterranean Fever (FMF) is the most common auto-inflammatory disease (prevalence: 1-5 / 10,000 inhabitants). It is due to mutations of the MEFV gene, encoding variants of the Pyrin inflammasome. Inflammasomes are protein complexes of innate immunity producing pro-inflammatory cytokines (interleukin-1β).

In vitro, preliminary results demonstrated that activation of the Pyrin inflammasome (measured by interleukin-1β concentration) by kinase inhibitors is significantly increased in FMF patients compared to subjects with a similar clinical picture, and healthy controls. In addition, a measure of cell death yielded significant results in differentiating patients from controls.

The investigators hypothesize that this fast and simple functional test can serve as a diagnostic tool for FMF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical picture compatible with an Familial Mediterranean Fever and an earlier genetic analysis finding a mutation of the MEFV gene;
* Newly diagnosed or undergoing follow-up (without criteria of delay or evolutionary stage);
* In the course of specific or non-specific treatment of the disease or without treatment;
* For whom a blood test is planned as part of the routine care;
* Of whom the informed non-opposition has been collected (parental authorization in the case of a minor patient);

Exclusion Criteria:

* patient under legal protection or under safeguard of justice or any other measures of protection (guardianship, curatorship);
* Person unable to express his consent;
* Person in emergency situation, vital or not;
* Infection known to HIV and / or HBV and / or HCV

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Familial Mediterranean Fever, patients controls with similar symptoms and healthy subjects who donated their blood to the French Blood Establishment.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Differences in interleukin-1bβ levels | Less than 48 hours
  Quantification of the capacity of interleukin-1β concentration measured in primary monocyte supernatants in response to kinase inhibitors, to discriminate Familial Mediterranean Fever subjects from control subjects (healthy subjects and subjects with symptoms similar to those of Familial Mediterranean Fever).
  Analysis have to be performed Less than 48 hours after blood sampling (only one sampling).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Service de néphrologie et rhumatologie pédiatrique, Hôpital Femme Mère Enfant, Bron
  - Unité Inserm U1111 & Service de Médecine Interne, Hôpital de la Croix-Rousse, Lyon
  - Service de Médecine Interne, Pavillon O - Hopital Edouard Herriot, Lyon
  - Service de Médecine Interne et pathologies vasculaires, Batiment 1B, Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: No